CLINICAL TRIAL: NCT04813965
Title: Downsides of Being Well-Informed: Tracking and Preventing Chemotherapy-Related Cognitive Problems in Breast Cancer Patients
Brief Title: Breast Cancer Patients' Cognitive Symptoms After Information About Chemotherapy-Related Cognitive Symptoms
Acronym: CONTEXT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: The Netherlands Cancer Institute (Other); St. Antonius Hospital (Other); Meander Medical Center (Other); Ziekenhuisgroep Twente (Other); Isala (Other); Deventer Ziekenhuis (Other); Rijnstate Hospital (Other); Franciscus Gasthuis (Other); St Jansdal Hospital (Other); UMC Utrecht (Other)
Responsible Party: Principal Investigator, Wendy Jacobs, MSc, study coordinator/PhD candidate, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: M13WEL; 2016-8178 (Other Grant/Funding Number: KWF Kankerbestrijding Nederland); 2011.WO34.C123 (Other Grant/Funding Number: Pink Ribbon Nederland); NL43939.031.13 (Registry Identifier: Registry ID: CCMO)
Record Dates: First submitted 2021-03-17; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer; Cognitive Symptoms; Cognitive Decline
Keywords: Breast cancer; Chemotherapy; Cognitive symptoms; Self-affirmation; Health communication; Nocebo; Stereotype threat
MeSH Terms: conditions — Breast Neoplasms; Neurobehavioral Manifestations; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: A multicenter, randomized, controlled, prospective, online survey study was conducted. Before completing the study's online baseline survey (pre-chemotherapy; T0), participants were randomly assigned by the online survey program to receive either: standard information on side-effects (control condition), or standard information with additional written information about chemotherapy-related cognitive symptoms (information condition), or standard and additional information with a subsequent self-affirmative text (information+SA condition; SA=self-affirmation). The online experimental texts were presented to patients once, directly after randomization at baseline. At six months (T1) and twelve months (T2) follow-up, all groups received identical general introductions and online surveys, without any experimental manipulations. Outside of the trial, all patients received treatment information from their medical oncologist according to local practice as part of their usual care.
Who Masked: Care Provider
Masking Description: Health care professionals were blinded to group assignment, but due to the nature of the study, patients were not. However, patients were not informed about the main outcomes and specific hypotheses of the study, or about the study's experimental conditions and the content of the texts that they did not receive until after T2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants in the control group received standard information on treatment side-effects.
- Information without self-affirmation (Experimental): Before completing the study's online baseline survey (pre-chemotherapy), participants in the information group received standard information with additional written information about potential chemotherapy-related cognitive symptoms.
  Interventions: Other: Written information about potential chemotherapy-related cognitive symptoms without self-affirmation
- Information with self-affirmation (Experimental): Before completing the study's online baseline survey (pre-chemotherapy), participants in the information+SA group (SA=self-affirmation) received standard and additional written information about potential chemotherapy-related cognitive symptoms with a subsequent self-affirmative text.
  Interventions: Other: Written information about potential chemotherapy-related cognitive symptoms with self-affirmation

INTERVENTIONS:
Other: Written information about potential chemotherapy-related cognitive symptoms without self-affirmation
  Other Names: Information
  Arms: Information without self-affirmation
Other: Written information about potential chemotherapy-related cognitive symptoms with self-affirmation
  Other Names: Information+SA
  Arms: Information with self-affirmation

SUMMARY:
Previous cross-sectional studies have shown that informing cancer patients about potential chemotherapy-related cognitive symptoms may negatively affect perceived cognitive symptoms and verbal memory performance. A multicenter, randomized study in newly diagnosed breast cancer patients receiving (neo) adjuvant chemotherapy was performed to evaluate this Adverse Information Effect (AIE) over time and investigated whether inviting patients to self-affirm can reduce such AIEs on perceived cognitive symptoms and cognitive test performance.

DETAILED DESCRIPTION:
Rationale:

Although information about their treatment and its side-effects is requested by cancer patients, is vital for informed decision making and can positively impact patients' health outcomes and illness perceptions, this kind of information can also adversely impact perceived cognitive symptoms and cognitive test performance. Previous studies have shown that informing cancer patients about potential chemotherapy-related cognitive symptoms may negatively affect perceived cognitive symptoms and verbal memory performance. A multicenter, randomized study in newly diagnosed breast cancer patients receiving (neo) adjuvant chemotherapy was performed to evaluate this Adverse Information Effect (AIE) over time and investigated whether inviting patients to self-affirm can reduce such AIEs on perceived cognitive symptoms and cognitive test performance.

Main objectives and hypotheses:

The overall aim of the study was to investigate the occurrence and duration of AIEs on the perceived frequency of cognitive symptoms, the perceived severity of cognitive symptoms and cognitive performance in breast cancer patients, and to examine ways to reduce such AIEs. First, evaluated the effect of providing breast cancer patients with additional factual written information about potential chemotherapy-related cognitive symptoms before chemotherapy-initiation on perceived cognitive symptoms and cognitive performance was evaluated, and the duration of such effects was assessed. Building on previous findings that breast cancer patients showed an increase in perceived cognitive symptoms and a decrease in verbal memory performance after receiving cognitive side-effect information, it was hypothesized that communicating about potential chemotherapy-related cognitive symptoms will result in AIEs, and it was explored to what extent these AIEs persist over time. Second, this study aimed to translate the beneficial effects of self-affirmation to the oncology domain, and examined the efficacy of a text-integrated self-affirmation intervention in reducing the impact of AIEs on perceived cognitive symptoms and cognitive performance in breast cancer patients when communicating about chemotherapy-related cognitive symptoms. It was hypothesized that a textual self-affirmation intervention would reduce AIEs in breast cancer patients, building on evidence from health promotion and stereotype threat research outside the oncology domain that individuals' self-concepts can be affirmed via text-integrated health messages and that allowing individuals the opportunity for self-affirmation can reduce stereotype threat effects.

The main research questions were:

1. Does written information about potential chemotherapy-related cognitive symptoms presented only once before treatment-initiation affect short- and longer-term perceived cognitive symptoms (the perceived frequency and severity of cognitive symptoms) and cognitive performance (verbal memory performance, information processing speed, executive functioning) in newly diagnosed breast cancer patients scheduled for (neo) adjuvant chemotherapy?
2. Does providing newly diagnosed breast cancer patients with a text integrated self-affirmation intervention after being informed about potential chemotherapy-related cognitive symptoms reduce AIEs on short- and longer-term perceived cognitive symptoms and cognitive performance?

Study procedure and outcome measures:

Before (neo) adjuvant chemotherapy, 160 newly diagnosed breast cancer patients were randomly allocated to receive either standard information on side-effects (control condition), or standard information with additional information about chemotherapy-related cognitive symptoms (information condition), or standard and additional information with a subsequent self-affirmative text (information+SA condition; SA=self-affirmation). Online-questionnaires were completed before chemotherapy (baseline, T0), 6-months (T1) and 12-months (T2) later to measure the perceived frequency (MOS-cog) and severity (MDASI-cog) of cognitive symptoms. Patients also completed two online neuro-psychological tests (Trail Making Test; TMT, and 15 Words test) to measure verbal memory performance, information processing speed and executive functioning. Additionally, several potential underlying mechanisms and risk factors of AIEs were examined, such as cancer related distress and performance worries. Baseline-to-follow-up analyses were performed using a mixed-effects modeling approach to compare groups over time.

ELIGIBILITY:
Inclusion Criteria:

* Primary breast cancer diagnosis stage I-III
* Scheduled to receive (neo) adjuvant chemotherapy
* 18 years or older
* Sufficient command of the Dutch language
* Internet access

Exclusion Criteria:

* A history of neurological and psychiatric symptoms that influence cognitive functioning
* Previous cancer diagnosis
* Using drugs
* Drinking more than three alcoholic drinks a day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2014-03-20 (Actual); Primary Completion 2016-09-23 (Actual); Study Completion 2016-09-23 (Actual)

PRIMARY OUTCOMES:
Between-group differences in mean change in the perceived frequency of cognitive symptoms from baseline to T1, and from baseline to T2. | Prior to chemotherapy-initiation (baseline; T0), six months (T1), and twelve months (T2) later
  Six items of the revised Medical Outcomes Study - cognitive functioning subscale (MOS-cog; Stewart & Ware, 1992) to measure the perceived frequency of cognitive symptoms. Participants indicated the frequency of experiencing a range of day-to-day problems in six aspects of cognitive functioning during the past week (including today). Higher mean scores indicate better perceived cognitive functioning (range 0-100).
Between-group differences in mean change in the perceived severity of cognitive symptoms from baseline to T1, and from baseline to T2. | Prior to chemotherapy-initiation (baseline; T0), six months (T1), and twelve months (T2) later
  Two items of the M.D. Anderson Symptom Inventory Multiple Myeloma module (MDASI-MM part 1; Cleeland et al., 2000; Jones et al., 2013) to measure the perceived severity of cognitive symptoms. Patients reported the severity of two cognitive symptoms at their worst in the last 24 hours on a 0-10 scale, with 0 being 'not present' and 10 being 'as bad as you can imagine': difficulty remembering and difficulty paying attention (concentrating). Higher mean scores indicate more severe symptoms.
Between-group differences in mean change in verbal memory performance from baseline to T1, and from baseline to T2. | Prior to chemotherapy-initiation (baseline; T0), six months (T1), and twelve months (T2) later
  Online, adapted version of the Groningen Fifteen Words Test (Rey, 1964) measuring immediate recall (range 0-45), delayed recall (range 0-15) and recognition (range 0-30). Higher scores indicate better performance.
Between-group differences in mean change in information processing speed and executive functioning from baseline to T1, and from baseline to T2. | Prior to chemotherapy-initiation (baseline; T0), six months (T1), and twelve months (T2) later
  Online version of the Trail Making Test (TMT; Reitan & Wolfson, 1985) part A and B (and TMT-B to TMT-A ratio B/A) to measure the speed of information processing and executive functioning. The score on each part represents the amount of time in seconds required to complete the task. Higher scores indicate worse information processing and executive functioning.

SECONDARY OUTCOMES:
Between-group differences in mean change in the levels of anxiety from baseline to T1, and from baseline to T2. | Prior to chemotherapy-initiation (baseline; T0), six months (T1), and twelve months (T2) later
  Dutch version of the Hospital Anxiety and Depression Scale (HADS; Spinhoven et al., 1997; Zigmond & Snaith, 1983) to measure levels of anxiety. Higher sum scores (range 0-21) indicate higher levels of anxiety.
Between-group differences in mean change in the levels of depression from baseline to T1, and from baseline to T2. | Prior to chemotherapy-initiation (baseline; T0), six months (T1), and twelve months (T2) later
  Dutch version of the Hospital Anxiety and Depression Scale (HADS; Spinhoven et al., 1997; Zigmond & Snaith, 1983) to measure levels of depression. Higher sum scores (range 0-21) indicate higher levels of depression.
Between-group differences in mean change in the perceived severity of other cancer-related symptoms from baseline to T1, and from baseline to T2. | Prior to chemotherapy-initiation (baseline; T0), six months (T1), and twelve months (T2) later
  Twelve items of the thirteen-item core M. D. Anderson Symptom Inventory (MDASI; part 1; Cleeland et al., 2000) to measure the perceived severity of other cancer-related symptoms. Participants reported the severity of twelve symptoms at their worst in the last 24 hours hours on a 0-10 scale, with 0 being 'not present' and 10 being 'as bad as you can imagine.' Difficulty remembering was excluded. Higher mean scores indicate more severe symptoms.
Between-group differences in pre-existing knowledge (prior to the experiment) about the potential cognitive symptoms of cancer treatment measured at twelve months follow-up (T2). | Measured at twelve months follow-up (T2)
  Participants indicated on one item (range 1-5) at the end of the T2 survey whether they had knowledge about the potential cognitive side-effects of cancer treatment prior to the experiment to measure pre-existing knowledge. Higher scores indicate more pre-existing knowledge.

OTHER OUTCOMES:
Between-group differences in mean change in the levels of the expected severity of cognitive symptoms from baseline to T1, and from baseline to T2. | Prior to chemotherapy-initiation (baseline; T0), six months (T1), and twelve months (T2) later
  An adapted version of two items of the M. D. Anderson Symptom Inventory Multiple Myeloma module (MDASI-MM; part 1; Cleeland et al., 2000; Jones et al., 2013) to measure the expected severity of cognitive symptoms during the next weeks (range 0-10). Higher scores indicate expectations of more severe cognitive symptoms.
Between-group differences in mean change in the levels of the expected severity of other cancer-related symptoms from baseline to T1, and from baseline to T2. | Prior to chemotherapy-initiation (baseline; T0), six months (T1), and twelve months (T2) later
  An adapted version of four items of the M. D. Anderson Symptom Inventory Multiple Myeloma module (MDASI-MM; part 1; Cleeland et al., 2000; Jones et al., 2013) to measure the expected severity of other cancer-related symptoms during the next weeks (range 0-10). Higher scores indicate expectations of more severe other cancer-related symptoms.
Between-group differences in mean change in the levels of motivation from baseline to T1, and from baseline to T2. | Prior to chemotherapy-initiation (baseline; T0), six months (T1), and twelve months (T2) later
  Five modified and translated items from the effort subscale of the Intrinsic Motivation Inventory (IMI; Ryan, 1982; Ryan & Deci, 2000) to measure the levels of motivation during the neuropsychological tasks (range 1-5). Higher mean scores indicate higher levels of motivation.
Between-group differences in mean change in the levels of worrying about cognitive test performance from baseline to T1, and from baseline to T2. | Prior to chemotherapy-initiation (baseline; T0), six months (T1), and twelve months (T2) later
  Four modified and translated items derived from the test anxiety subscale of the Motivated Strategies for learning Questionnaire (Pintrich & De Groot, 1990) to measure the levels of worrying about cognitive test performance (range 1-5). Higher mean scores denote higher levels of worries.
Low cancer-specific distress versus high cancer-specific distress subgroup analysis. | Prior to chemotherapy-initiation (baseline; T0), six months (T1), and twelve months (T2) later
  Seven items of the intrusion subscale of the Dutch version of the Impact of Events Scale (Horowitz, Wilner, & Alvarez, 1979; Van der Ploeg et al., 2004) to assess the levels of intrusion of cancer related stressful thoughts (range 0-28). Higher sum scores indicate higher intrusion when confronted with the stressful experience of being treated for cancer.
Low stigma consciousness versus high stigma consciousness subgroup analysis. | Prior to chemotherapy-initiation (baseline; T0), six months (T1), and twelve months (T2) later
  Eight translated and adapted items derived from the 10-item Stigma Consciousness Questionnaire to measure the extent to which patients expect to be stereotyped by others (Brown & Pinel, 2003; cf. Jacobs, Das, & Schagen, 2017; range 1-5). Higher mean scores indicate higher levels of stigma consciousness.
Low domain identification versus high domain identification subgroup analysis. | Prior to chemotherapy-initiation (baseline; T0), six months (T1), and twelve months (T2) later
  Three adapted and translated items from the math identification subscale of the Social Identities and Attitudes Scale (SIAS; Picho & Brown, 2011), to measure the extent to which participants identify with the domain of 'cognition' and the level of importance of their cognition (range 1-5). Higher mean scores indicate higher levels of domain identification.
Low group identification versus high group identification subgroup analysis. | Prior to chemotherapy-initiation (baseline; T0), six months (T1), and twelve months (T2) later
  Two newly developed items and four items derived and adapted from Doosje and colleagues (Doosje, Ellemers, & Spears, 1995), Spears and colleagues (Spears, Doosje, & Ellemers, 1997), and Quayle (2011) to measure the level of group identification, that is to what extent participants identify with other (ex) cancer patients (range 1-5). Higher mean scores indicate higher levels of group identification.
Low information monitoring versus high information monitoring subgroup analysis. | Prior to chemotherapy-initiation (baseline; T0), six months (T1), and twelve months (T2) later
  Information monitoring was measured by one item that asked patients how often during the past weeks they searched for health- and cancer related information (range 0-4). Higher scores indicate higher levels of information monitoring.
Between-group differences in changes in information source from baseline to T1, and from baseline to T2. | Prior to chemotherapy-initiation (baseline; T0), six months (T1), and twelve months (T2) later
  One item to indicate which information sources participants used (twelve options; for example information leaflets yes/no).
Between-group differences in changes in information content from baseline to T1, and from baseline to T2. | Prior to chemotherapy-initiation (baseline; T0), six months (T1), and twelve months (T2) later
  One item to assess what information content participants looked for (six options; for example information about chemotherapy side-effects yes/no).
Between-group differences in stereotype self-relevance measured at twelve months follow-up (T2). | Measured at twelve months follow-up (T2)
  At twelve months follow-up (T2), stereotype self-relevance was measured using one item that assessed perceived self-relevance of the chemotherapy-impairs-cognition stereotype: 'To what extent does the phenomena 'Chemo brain' apply to you?' (range 1-5). Higher scores indicate higher levels of self-relevance.
Between-group differences in the extent to which participants attributed their own and others' cognitive symptoms to chemotherapy measured at twelve months follow-up (T2). | Measured at twelve months follow-up (T2)
  At twelve months follow-up (T2), two items asked participants to indicate the extent to which they attributed their own and others' cognitive symptoms to chemotherapy (range 1-5). Higher scores indicate higher levels of attribution of cognitive symptoms to chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Enny Das, PhD, Principal Investigator — Radboud University Medical Center; Sanne B Schagen, PhD, Principal Investigator — The Netherlands Cancer Institute; Gabe S Sonke, PhD, MD, Principal Investigator — The Netherlands Cancer Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jacobs W, Schagen SB, Brouwer SM, Kieffer JM, Baas IO, Los M, Sonke GS, Das E. The Effects of Being Informed About Chemotherapy-Related Cognitive Symptoms With And Without Self-Affirmation on Perceived Cognitive Symptoms of Breast Cancer Patients: A Randomized Prospective, Longitudinal Study. Clin Breast Cancer. 2022 Jul;22(5):439-454. doi: 10.1016/j.clbc.2022.03.001. Epub 2022 Mar 26. PMID 35491320